CLINICAL TRIAL: NCT01504698
Title: Manipulative Treatment of Children With Neck and Back Pain. A Randomised Controlled Trial of 1200 Children From 3rd to 7th Grade
Brief Title: Manipulative Treatment of Children With Neck and Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Chiropractors Fund (Unknown); Municipality of Svendborg (Unknown); Nordic Institute of Chiropractic and Clinical Biomechanics (Other); Sygehus Lillebaelt (Other); IMK Foundation (Unknown); Chiroform (Unknown)
Responsible Party: Principal Investigator, Kristina Boe Dissing, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVKS-20110042
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Neck Pain; Back Pain
Keywords: Manipulative treatment; Children; Neck pain; Back pain; Effect; Adolescence; Advise; Exercise
MeSH Terms: conditions — Neck Pain; Back Pain; Motor Activity | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with manipulation (Experimental)
  Interventions: Procedure: Advice and exercise-based treatment plus joint manipulation
- Treatment without manipulation (Active Comparator)
  Interventions: Procedure: Advice and exercise-based treatment

INTERVENTIONS:
Procedure: Advice and exercise-based treatment plus joint manipulation — The treatment can consist of advice, activation and exercise and/or manual soft-tissue treatment plus joint manipulation.The areas and frequency of manipulative treatment will be determined by the chiropractor and will consist of high-velocity, low-amplitude manipulation and/or mobilization to the spine and/or the extremities.
  Arms: Treatment with manipulation
Procedure: Advice and exercise-based treatment — The treatment can consist of advice, activation and exercise and/or manual soft-tissue treatment. However, assisted stretching is not allowed as this will approach mobilization.
  Arms: Treatment without manipulation

SUMMARY:
The purpose of this study is to determine the effect of manipulative treatment of children with neck and back pain. Because manipulation is the most frequently used treatment of musculoskeletal complaints in children, and an increasing number of Danish children see a chiropractor, it appears obvious to start the search for evidence by examining the effect of this treatment.

DETAILED DESCRIPTION:
Parents receive text messages [SMS) on a weekly basis inquiring about the child's musculoskeletal pain as well as amount and types of sport during leisure time the past week. Following a report of pain, the parents will be interviewed by phone by a member of the clinical team, consisting of two licensed physical therapists and two licensed chiropractors, for a thorough description of the complaint. Based on this, the interviewer determines whether the complaint is negligible or whether the child should be seen by a member of the clinical team, in which case the child will be examined at his or her school. At this examination, the child will be evaluated for inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Pain in neck or back equal to or greater than 3 on an 11-box numerical rating scale for more than three days.

Exclusion Criteria:

* If a serious pathology or injury is suspected, the child will be referred to a secondary care sports injury center for diagnostic work-up and/or imaging.
* Handicaps which prevents normal physical activity.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of recurrences during the follow-up period. | 2 1/2 year
  Weekly reports of pain by sms

SECONDARY OUTCOMES:
Global perceived effect after two weeks | 2 weeks
  Questionnaire
Change in pain intensity (Numerical Rating Scale) | After one and two weeks
  Questionnaire
Average duration of complaint time for each episode | Up till 2 1/2 years
  Weekly reports of pain by sms
Total duration of complaint time during the follow-up period (combination of duration and recurrences) | 2 1/2 year

CONTACTS AND LOCATIONS:
Overall Officials: Niels Wedderkopp, Ph.D., Study Director — University of Southern Denmark
Locations (1):
- 13 Municipal Schools, Svendborg, Denmark

REFERENCES:
- [Derived] Dissing KB, Vach W, Hartvigsen J, Wedderkopp N, Hestbaek L. Potential treatment effect modifiers for manipulative therapy for children complaining of spinal pain.Secondary analyses of a randomised controlled trial. Chiropr Man Therap. 2019 Dec 10;27:59. doi: 10.1186/s12998-019-0282-7. eCollection 2019. PMID 31827767
- [Derived] Dissing KB, Hartvigsen J, Wedderkopp N, Hestbaek L. Conservative care with or without manipulative therapy in the management of back and/or neck pain in Danish children aged 9-15: a randomised controlled trial nested in a school-based cohort. BMJ Open. 2018 Sep 10;8(9):e021358. doi: 10.1136/bmjopen-2017-021358. PMID 30206079
- [Derived] Dissing KB, Hartvigsen J, Wedderkopp N, Hestbaek L. Conservative care with or without manipulative therapy in the management of back and neck pain in Danish children aged 9-15. Study protocol for a randomized controlled trial. Chiropr Man Therap. 2016 Jan 28;24:5. doi: 10.1186/s12998-016-0086-y. eCollection 2016. PMID 26823970